CLINICAL TRIAL: NCT05934045
Title: Deciphering the Role of Circular RNAs in the Pathogenesis and Therapy Resistance of ALKpositive Anaplastic Large-cell Lymphoma
Brief Title: Deciphering the Role of Circular RNAs in ALKpositive Anaplastic Large-cell Lymphoma
Acronym: CIRComa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0507; French Ministry of Health (Other Grant/Funding Number: PRT-K22-051)
Record Dates: First submitted 2023-06-23; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: ALK-Positive Anaplastic Large Cell Lymphoma
Keywords: cancer
MeSH Terms: conditions — Neoplasms | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALCL patient samples (serum): serum collected at diagnosis, during treatment and/or at relapse
  Interventions: Biological: RNAseq

INTERVENTIONS:
Biological: RNAseq — there is no intervention done.

SUMMARY:
The objective of thE project is to determine, whether circRNAs could be used as circulating prognostic and/or predictive biomarkers of ALK+ ALCL resistance to treatment and whether they can be exploited as therapeutic targets.

DETAILED DESCRIPTION:
Anaplastic large-cell lymphoma (ALCL) is an aggressive T-cell pediatric lymphoma. 85% of ALK+ ALCL cases harbor a fusion between the nucleophosmin (NPM) and anaplastic lymphoma kinase (ALK) genes, leading to a constitutively activated and oncogenic fusion protein. Most ALK+ ALCL cases initially respond well to the frontline chemotherapy, but 30% of patients relapse and are of poor prognosis. Understanding the origins of therapy resistance is of major importance to improve treatment and patient prognosis. Current research highlights deregulated expression of regulatory non-coding RNAs (ncRNAs) as an important factor in therapy resistance. To date, microRNAs and long noncoding RNAs have been linked to therapy resistance in ALK+ ALCL. Circular RNAs (circRNAs) are a class of highly stable noncoding RNAs that have recently come into the focus of researchers. circRNAs can control target gene expression by e.g. interacting with microRNAs or proteins. This project aims to elucidate their role in ALK+ ALCL biology including their impact on noncoding RNA networks and therapy resistance. This project will (1) identify a signature of circRNAs associated with therapy resistance in ALK+ ALCL, (2) analyze their effect on treatment response, (3) elucidate their mechanism of action, and (4) evaluate circRNA candidates as predictive and prognostic plasma biomarkers using liquid biopsies. The goal of the study is to characterize the role of candidate circRNAs in this well-defined cancer type, which can serve as a model for other ALK+ cancers. Project results will add to the current mechanistic understanding of ALK+ ALCL pathogenesis and the origins of therapy resistance, and could define new druggable targets and associated predictive biomarkers for high-risk disease. Establishing the blood-based alternative confirmation for the ALK+ ALCL diagnosis could also produce a less invasive predictive tool capable of longitudinal patient monitoring for early relapse detection.

ELIGIBILITY:
Inclusion Criteria:

* patient at diagnosis of ALK+ ALCL
* patient at the time of relapse for ALK+ ALCL
* patient without ALK+ ALCL

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient at diagnosis of ALK+ ALCL, patient at the time of relapse for ALK+ ALCL, patient without ALK+ ALCL
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with relapse and circulating circRNA | 1 year after the end of treatment
  RNAseq analysis

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Lamant, Principal Investigator — University Hospital, Toulouse
Locations (1):
- IUCT-Oncopole University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No